CLINICAL TRIAL: NCT00006243
Title: Melanoma Vaccines: Differentiation Antigen Peptides (MART-1:27-35, Tyrosinase and Gp-100) as Immune Targets
Brief Title: Vaccine Therapy and Sargramostim in Treating Patients With Stage IV Malignant Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02359; MC9973; CDR0000068171 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-09-11; First posted 2003-05-22 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — gp100 Melanoma Antigen; incomplete Freund's adjuvant; montanide ISA 51; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

ARMS (3):
- Arm I (vaccine therapy) (Experimental): Patients receive tyrosinase peptide, MART-1:27-35 peptide vaccine, and gp100 antigen admixed in incomplete Freund's adjuvant SC on day 1 of weeks 0, 3, 6, 9, 12, and 24.
  Interventions: Biological: tyrosinase peptide; Biological: MART-1:27-35 peptide vaccine; Biological: gp100 antigen; Biological: incomplete Freund's adjuvant; Other: laboratory biomarker analysis
- Arm II (vaccine therapy and lower-dose sargramostim) (Experimental): Patients receive tyrosinase peptide, MART-1:27-35 peptide vaccine, and gp100 antigen admixed in incomplete Freund's adjuvant SC and lower-dose sargramostim SC on day 1 of weeks 0, 3, 6, 9, 12, and 24.
  Interventions: Biological: tyrosinase peptide; Biological: MART-1:27-35 peptide vaccine; Biological: gp100 antigen; Biological: incomplete Freund's adjuvant; Biological: sargramostim; Other: laboratory biomarker analysis
- Arm III (vaccine therapy and higher-dose sargramostim) (Experimental): Patients receive tyrosinase peptide, MART-1:27-35 peptide vaccine, and gp100 antigen admixed in incomplete Freund's adjuvant SC and higher-dose sargramostim SC on day 1 of weeks 0, 3, 6, 9, 12, and 24.
  Interventions: Biological: tyrosinase peptide; Biological: MART-1:27-35 peptide vaccine; Biological: gp100 antigen; Biological: incomplete Freund's adjuvant; Biological: sargramostim; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: tyrosinase peptide — Given SC
  Other Names: TYRP
Biological: MART-1:27-35 peptide vaccine — Given SC
Biological: gp100 antigen — Given SC
  Other Names: gp100
Biological: incomplete Freund's adjuvant — Given SC
  Other Names: IFA; ISA-51; Montanide ISA 51
Biological: sargramostim — Given SC
  Other Names: GM-CSF; Leukine; Prokine
  Arms: Arm II (vaccine therapy and lower-dose sargramostim); Arm III (vaccine therapy and higher-dose sargramostim)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized pilot clinical trial studies vaccine therapy and sargramostim in treating patients with stage IV malignant melanoma. Vaccines made from melanoma peptides or antigens may help the body build an effective immune response to kill tumor cells. Colony-stimulating factors, such as sargramostim, increase the number of white blood cells and platelets found in bone marrow or peripheral blood. Giving vaccine therapy together with sargramostim may be an effective treatment for malignant melanoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the immunological effects of immunization protocols utilizing MART-1:27-35 (MART-1:27-35 peptide vaccine), tyrosinase (tyrosinase peptide) or gp-100 (gp100 antigen) peptides suspended in incomplete Freund's adjuvant (IFA) in the presence of two different concentrations of sargramostim (GM-CSF).

II. Define the safety and toxicity profile of an immunization protocol utilizing varying concentrations of MART-1:27-35, tyrosinase and gp-100 peptides suspended in IFA in the presence of two different concentrations of GM-CSF.

III. Collect preliminary data on therapeutic efficacy as it relates to parameters of immune function in patients with stage IV malignant melanoma.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive tyrosinase peptide, MART-1:27-35 peptide vaccine, and gp100 antigen admixed in incomplete Freund's adjuvant subcutaneously (SC) on day 1 of weeks 0, 3, 6, 9, 12, and 24.

ARM II: Patients receive tyrosinase peptide, MART-1:27-35 peptide vaccine, and gp100 antigen admixed in incomplete Freund's adjuvant SC and lower-dose sargramostim SC on day 1 of weeks 0, 3, 6, 9, 12, and 24.

ARM III: Patients receive tyrosinase peptide, MART-1:27-35 peptide vaccine, and gp100 antigen admixed in incomplete Freund's adjuvant SC and higher-dose sargramostim SC on day 1 of weeks 0, 3, 6, 9, 12, and 24.

In all arms, treatment may repeat every 3 months for up to 18 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Human leukocyte antigen (HLA)-A2 positive
* Histologic proof of stage IV malignant melanoma with measurable disease
* Absolute neutrophil count (ANC) >= 1500
* Platelets (PLT) >= 100,000
* Alkaline phosphatase (Alk phos) =< 3 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) =< 3 x ULN
* Creatinine (Creat) =< 1.5 x ULN
* Hemoglobin (Hgb) > 9.0
* Ability to provide informed consent
* Willingness to return to a Mayo Clinic institution for follow-up
* Life expectancy >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2

Exclusion Criteria:

* Uncontrolled or current infection
* Prior immunization with differentiation antigen peptides
* Known standard therapy for the patient's disease that is potentially curative or proven capable of extending life expectancy
* Any of the following prior therapies:

  * Chemotherapy =< 4 weeks
  * Mitomycin C/nitrosoureas =< 6 weeks
  * Immunotherapy =<4 weeks
  * Biologic therapy =< 4 weeks
  * Radiation therapy =< 4 weeks
  * Radiation to > 25% of bone marrow
* Failure to fully recover from effects of prior chemotherapy regardless of interval since last treatment
* New York Heart Association classification III or IV
* Seizure disorder
* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.)
* Other concurrent chemotherapy, immunotherapy, or radiotherapy
* Active psychiatric disorder requiring medications (anti-psychotics)
* Known central nervous system metastases or carcinomatous meningitis
* History of other malignancy in last 5 years with the exception of basal cell or squamous cell carcinoma of the skin treated with local resection only (it is impossible to predict the effect of study treatment on other, potentially dormant malignant diseases)
* Known immune deficiency (patients with known immune deficiencies will likely not be able to mount an immune response to the study vaccine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2000-10; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Changes in tumor antigen peptide specific immune responses | Baseline and 24 weeks
  Plots of the percent changes in these factors from their pretreatment levels against time will be constructed.

SECONDARY OUTCOMES:
Number and severity of hematologic and non-hematologic toxicities observed using the Common Toxicity Criteria (CTC) version 2.0 | Up to 3 years
Proportion of objective responses (complete response [CR] and partial response [PR]) observed | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States